CLINICAL TRIAL: NCT07187791
Title: Validation of CT KUB in Assesment of Renal Cysts
Brief Title: CT KUB in Renal Cysts
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Thomas Nabeel Mikha Saied, Resident Doctor, Assiut University
Other Study IDs: CT in Renal cysts
Record Dates: First submitted 2025-09-10; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: CT KUB; Renal Cyst
MeSH Terms: interventions — Tomography, X-Ray Computed; Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CT scan — All Patients will undergo CT KUB cyst evaluation Qualitatively regarding Gross Picture in Imaging and Quantitavely using Hausfield units then patients will undergo Abdomianl ultrasound
  Other Names: Ultrasound

SUMMARY:
1. Primary (main):

   1. Determine the diagnostic accuracy of CT KUB in differentiating between benign and suspicious renal cysts according to the Bosniak classification.
2. Secondary (subsidiary):

   1. Assess interobserver agreement in CT KUB interpretation among radiologists with varying levels of expertise.
   2. Identify limitations and pitfalls in the use of non-contrast CT KUB for characterizing renal cysts.

DETAILED DESCRIPTION:
Renal cysts are among the most frequently encountered incidental findings(1) on abdominal imaging, particularly with the increasing use of cross-sectional imaging. Most simple cysts are benign and require no further evaluation.

However, complex cystic lesions pose a diagnostic challenge, necessitating accurate characterization to distinguish benign from malignant lesions.(2).

While CT KUB is highly effective for detecting urinary tract stones, there are several limitations and pitfalls we should be aware of as Limited Soft Tissue Assessment as without contrast, masses, infections, or vascular lesions may not be clearly visible also some tumors called isodensity tumors, have similar intensity values to the surrounding normal tissues.(3).

Segmentation of kidney tumors on CT KUB images adds challenges compared to contrast-enhanced CT (CECT) images, due to low contrast and lack of multiphase images. On CECT images, the kidney tumors have different intensity values compared to the normal tissues.(4).

Validating CT KUB's accuracy in assessing renal cysts could have significant implications for clinical decision making, especially in resource-limited or urgent care settings

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for CT KUB with detectable Renal cysts

Exclusion Criteria:

* 1-Patients with known renal tumors.
* 2-Inadequate imaging quality: CT KUB with severe motion/streak artifact or incomplete anatomical coverage preventing lesion assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Renal Cysts referred to CT KUB for any indication
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Validiation of CT KUB results in assesment of Renal Cystic Lesions prospectively in comparison to Ultrasonographic as in terms of Sensitivity and Specificity regarding evalution of Cystic lesion complexity according to Bosniak Classification | From Time of CT KUB referal till accurate diagnosis of Cystic lesion up to 24 weeks
  CT KUB cyst evaluation Qualitatively as Gross Picture and Quantitavely using Hausfield units then Abdomianl ultrasound , otherwise Bosniak I Renal cysts will undergo further assessment contrast-enhanced CT then Follow Up or Histopathology Data will be captured on a pre-piloted electronic case report form with de-identified study codes. Statistical analysis (sensitivity, specificity, PPV, NPV, accuracy, ROC/AUC) and inter-/intra-observer agreement (κ/ICC) will be conducted using SPSS/R/Stata. Quality assurance will follow institutional scanner QA logs, a priori reader calibration, and an audit-trailed database.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forookhi, A., Bicchetti, M., Lucciola, S. et al. The thin line that made the difference: a case report on a Bosniak IIF renal cystic mass treated with cyst decortication. Egypt J Radiol Nucl Med 53, 115 (2022). https://doi.org/10.1186/s43055-022-00791-3
- [Background] Smith AD, Remer EM, Cox KL, Lieber ML, Allen BC, Shah SN, Herts BR. Bosniak category IIF and III cystic renal lesions: outcomes and associations. Radiology. 2012 Jan;262(1):152-60. doi: 10.1148/radiol.11110888. Epub 2011 Nov 21. PMID 22106359